CLINICAL TRIAL: NCT04816422
Title: Proprioceptive Neuromuscular Facilitation (PNF) Techniques to Improve Bed Mobility, Transfer and Early Trunk Control in Stroke Patients
Brief Title: PNF Techniques to Improve Bed Mobility, Transfer and Early Trunk Control in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/19/1011 Naeem Abbas
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive neuromuscular facilitation (Experimental): Bilateral upper extremity pattern for trunk by Chopping, Lifting 2. Bilateral lower extremity pattern for trunk. 3. Trunk lateral flexion. 4. Combination patterns for the trunk by Upper and lower trunk flexion, Upper trunk flexion with lower trunk extension, Upper and lower trunk extension, Upper trunk extension with lower trunk flexion.
  Interventions: Other: Proprioceptive neuromuscular facilitation
- Conventional treatment (Active Comparator): Procedure Group 2 has received conventional trunk exercise program for 45 min/day, 4 days
  / week for the period of 4 weeks the intervention includes static and dynamic functional trunk movement and strengthening exercise to the trunk muscles which includes motor developmental patterns, basic trunk movement, trunk-arm linked movements, trunk-leg linked patterns in sitting, transfer activities, with 2 minutes rest in between the repetition of each set, Progression will be made by increasing the repetition and resistance According to individual ability.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation — rocedure
  1. Bilateral upper extremity pattern for trunk by Chopping, Lifting
  2. Bilateral lower extremity pattern for trunk.
  3. Trunk lateral flexion.
  4. Combination patterns for the trunk by Upper and lower trunk flexion, Upper trunk flexion with lower trunk extension, Upper and lower trunk extension, Upper trunk extension with lower trunk flexion.
  Arms: Proprioceptive neuromuscular facilitation
Other: Conventional treatment — Group 2 has received conventional trunk exercise program for 45 min/day, 4 days
  / week for the period of 4 weeks the intervention includes static and dynamic functional trunk movement and strengthening exercise to the trunk muscles which includes motor developmental patterns, basic trunk movement, trunk-arm linked movements, trunk-leg linked patterns in sitting, transfer activities, with 2 minutes rest in between the repetition of each set, Progression will be made by increasing the repetition and resistance According to individual ability.
  Arms: Conventional treatment

SUMMARY:
Trunk control is an important factor which is disturbed after the stroke. The literature reviews suggest that trunk exercises are required to achieve good trunk stability which is essential for balance, daily functional activities and higher function tasks. By keeping these facts in view present study aims at evaluating the efficacy of PNF techniques & conventional trunk exercise to improve trunk control in recovery stage hemiplegic patients Objective: To determine Proprioceptive neuromuscular facilitation (PNF) Techniques to improve bed mobility, transfer and early trunk control in Stroke patients

DETAILED DESCRIPTION:
50 patients was included and allocated into 2 groups, group A consisting of 25 patients who received PNF techniques for trunk to improve trunk control. Group B consisting of 25 patients who received conventional trunk exercises to improve trunk control. Trunk control was assessed pre and post treatment with the help of Trunk Impairment Scale and ICU mobility scale. Data was collected by ICU mobility scale & Trunk impairment scale

ELIGIBILITY:
Inclusion Criteria:

* Stroke (Acute stage)
* First attack without any prior residual impairment.
* Middle Cerebral Artery syndrome

Exclusion Criteria:

* Cognitive deficits or aphasia
* Neurological disorders e.g, Parkinson's disease.
* Heart failure
* Systemic orthopaedic and psychological disorders

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
ICU mobility scale | 2 months
  The ICU Mobility Scale (IMS) is an 11-item categorical scale that measures the highest level of functional mobility of patients within the intensive care unit (ICU) setting.
Trunk impairment scale | 2 months
  To examine the clinimetric characteristics of the Trunk Impairment Scale (TIS). This newly developed scale evaluates motor impairment of the trunk after stroke. The TIS scores, on a range from 0 to 23, static and dynamic sitting balance as well as trunk co-ordination. It also aims to score the quality of trunk movement and to be a guide for treatment

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Binash afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guiu-Tula FX, Cabanas-Valdes R, Sitja-Rabert M, Urrutia G, Gomara-Toldra N. The Efficacy of the proprioceptive neuromuscular facilitation (PNF) approach in stroke rehabilitation to improve basic activities of daily living and quality of life: a systematic review and meta-analysis protocol. BMJ Open. 2017 Dec 12;7(12):e016739. doi: 10.1136/bmjopen-2017-016739. PMID 29233831
- [Background] Li F, Sun Q, Shao XM, Xie JJ, Liu HB, Xu Y, Yang WD. [Electroacupuncture combined with PNF on proprioception and motor function of lower limbs in stroke patients: a randomized controlled trial]. Zhongguo Zhen Jiu. 2019 Oct 12;39(10):1034-40. doi: 10.13703/j.0255-2930.2019.10.002. Chinese. PMID 31621252
- [Background] Krukowska J, Bugajski M, Sienkiewicz M, Czernicki J. The influence of NDT-Bobath and PNF methods on the field support and total path length measure foot pressure (COP) in patients after stroke. Neurol Neurochir Pol. 2016 Nov-Dec;50(6):449-454. doi: 10.1016/j.pjnns.2016.08.004. Epub 2016 Aug 20. PMID 27585746
- [Background] Sharma V, Kaur J. Effect of core strengthening with pelvic proprioceptive neuromuscular facilitation on trunk, balance, gait, and function in chronic stroke. J Exerc Rehabil. 2017 Apr 30;13(2):200-205. doi: 10.12965/jer.1734892.446. eCollection 2017 Apr. PMID 28503533
- [Background] Junior VADS, Santos MS, Ribeiro NMDS, Maldonado IL. Combining Proprioceptive Neuromuscular Facilitation and Virtual Reality for Improving Sensorimotor Function in Stroke Survivors: A Randomized Clinical Trial. J Cent Nerv Syst Dis. 2019 Jul 25;11:1179573519863826. doi: 10.1177/1179573519863826. eCollection 2019. PMID 31384139
- [Background] Kim BR, Kang TW. The effects of proprioceptive neuromuscular facilitation lower-leg taping and treadmill training on mobility in patients with stroke. Int J Rehabil Res. 2018 Dec;41(4):343-348. doi: 10.1097/MRR.0000000000000309. PMID 30067555
- [Background] Shim J, Hwang S, Ki K, Woo Y. Effects of EMG-triggered FES during trunk pattern in PNF on balance and gait performance in persons with stroke. Restor Neurol Neurosci. 2020;38(2):141-150. doi: 10.3233/RNN-190944. PMID 32250337
- [Background] Smedes F, Giacometti da Silva L. Motor learning with the PNF-concept, an alternative to constrained induced movement therapy in a patient after a stroke; a case report. J Bodyw Mov Ther. 2019 Jul;23(3):622-627. doi: 10.1016/j.jbmt.2018.05.003. Epub 2018 May 31. PMID 31563380
- [Background] Cayco CS, Gorgon EJR, Lazaro RT. Effects of proprioceptive neuromuscular facilitation on balance, strength, and mobility of an older adult with chronic stroke: A case report. J Bodyw Mov Ther. 2017 Oct;21(4):767-774. doi: 10.1016/j.jbmt.2016.10.008. Epub 2016 Oct 27. PMID 29037625